CLINICAL TRIAL: NCT03987360
Title: Educational and Cultural Engagement and Incidence of Health Adverse Events: Results From the Canadian Longitudinal Study on Aging
Brief Title: Educational and Cultural Engagement and Incidence of Health Adverse Events
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-1842
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Older Adults; Depression; Cognitive Decline
MeSH Terms: conditions — Depression; Cognitive Dysfunction | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Participants who attended different educational and cultural activities either in a community centers or public institutions like arts museums or universities.

SUMMARY:
This study evaluated if the social and cultural activities decrease the incidence of dementia and frailty conditions.

DETAILED DESCRIPTION:
The past decade has been characterized by the involvement of Museums in individual health prevention and promotion by using art-based activities to improve quality of life and well-being. Visiting museum or over cultural and educational activity could be used for health prevention and promotion. For the development of appropriate educational and cultural activities, there is a need, first, to improve knowledge about social and health condition of older adult, and second to examine the effects of engagement in educational and social activity on incidence of health adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Being 50 years and over
* Being enrolled in the Canadian Longitudinal Study on Aging
* Actively involved in social and cultural activities

Exclusion Criteria:

* Never enrolled in the Canadian Longitudinal Study on Aging
* Less than 50 years old

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People from Canada who participate in the Canadian Longitudinal Study on Aging. Participants who have the habits to go to museums for art classes, workshops, guided visits, and others arts activities. Participants of Canadian Longitudinal Study on Aging who are involved in art and educational activities in their communities.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2020-03-31 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Depression | around 20 years
  It will be used the Depression scale which has a score of 10 or less. Each participant will be asses based on this scale. The depression scale evaluates the depression symptoms for a time period.

SECONDARY OUTCOMES:
Motoric cognitive risk syndrome | around 20 years
  Motoric cognitive risk syndrome represents a pre-dementia syndrome characterized by cognitive complaints and a slow gait speed.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada